CLINICAL TRIAL: NCT00686816
Title: A Study Among Pre-diabetic, Obese Women to Evaluate the Weight Loss Effects of a Non-Digestible Fat Substitute
Brief Title: Weight Loss in Pre-diabetic, Obese Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Muhammad Rehman, MD, Procter & Gamble
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008030
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
Keywords: pre-diabetic; obese
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — Caloric Restriction; sucrose polyester

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Low calorie diet
- 2 (Experimental)
  Interventions: Dietary Supplement: Olestra

INTERVENTIONS:
Dietary Supplement: Low calorie diet — low calorie diet
  Arms: 1
Dietary Supplement: Olestra — low calorie Olestra diet
  Arms: 2

SUMMARY:
This is a six (6) month, single center, randomized, double-blind, parallel, controlled-feeding weight-loss study comparing two dietary groups (triglyceride and olestra) in pre-diabetic obese women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal
* BMI 30-45 kg/meter squared
* waist circumference greater than 88 cm
* blood glucose level 5.8-6.9 mmol/l

Exclusion Criteria:

* Pre-diabetic
* pregnant
* nursing
* food preferences not compatible with the study diet
* allergies or food sensitivities with any of the study diet

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
weight loss | 3 months

SECONDARY OUTCOMES:
Weight maintained | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, MD, Principal Investigator — Russian Institue of Nutrition
Locations (1):
- Vasily Isakov, MD, Moscow, Russia